CLINICAL TRIAL: NCT01702961
Title: A Current Practice Study of Rituxan in Patient Receiving BEAM Chemotherapy and Autologous Blood Stem Cell Transplantation for High Risk Lymphoma or Hodgkin's Disease
Brief Title: Rituxan + BEAM and Auto Stem Cell Transplant for High Risk Lymphoma or Hodgkin's Disease
Acronym: Rituxan+BEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, George Carrum, Associate Professor; Director-Adult Outpatient Clinic, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-11892; Rituxan+BEAM (Other: BCM Center for Cell and Gene Therapy)
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma; Hodgkin's Disease
Keywords: Lymphoma; Hodgkin's Disease
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Melphalan; Cytarabine; Etoposide; Carmustine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BEAM+R: Autologous Stem Cell Transplant (Other): Ara-C, VP-16, BCNU, Melphalan, Rituxan and Stem Cells
  Interventions: Drug: Melphalan; Drug: Ara-C; Drug: VP-16; Drug: BCNU; Drug: Rituxan; Drug: Stem Cells

INTERVENTIONS:
Drug: Melphalan — Given on Day -1
  Melphalan is administered according to the current SOP.
  Other Names: Alkeran
Drug: Ara-C — 200 mg/m2 IB BID given on Days -5, -4, -3, -2
  Other Names: Cytarabine; Cytosar-u
Drug: VP-16 — 200 mg/m2 IV BID given on Days -5, -4, -3, -2
  Other Names: Etoposide
Drug: BCNU — BCNU 300 mg/m2 IV given on Day -6
  Other Names: Carmustine
Drug: Rituxan — 375 mg/m2 IB given on Days -6, +14, +21, +28
  Other Names: Rituxamib
Drug: Stem Cells — Stem cells given on Day 0
  Other Names: Autologous Blood Stem Cells

SUMMARY:
High-dose chemotherapy followed by autologous (the patient's own) peripheral blood (circulating blood) stem cell (cells that divide to form white cells, red cells and cells that help clot) transplantation is a conventional treatment for patients with lymphoma (cancer of lymph glands) and Hodgkin's disease (cancer of lymph glands) after first relapse (recurrence of disease). For patients who did not have a complete response after traditional chemotherapy, the chance is high that the tumor will return even after high-dose chemotherapy. To improve the response and decrease the chance of relapse, doctors have used rituximab, an antibody that kills lymphoma cells, both before and after transplantation. These doctors have reported that more patients had control of the tumor for an extended period of time using rituximab with high-dose chemotherapy with autologous stem cell transplantation. How widely this is applicable is not known.

The purpose of this clinical research trial is to confirm that there is a good control of tumor in patients with lymphoma or Hodgkin's disease treated with rituximab and conventional stem cell transplantation.

DETAILED DESCRIPTION:
Subjects will receive the chemotherapy through a plastic tube (catheter) placed into a vein under the collarbone. The antibody rituximab is given on the day of admission. The subject will also start a six-day course of chemotherapy at that time. The chemotherapy will consist of the following drugs: BCNU, etoposide also called VP-16, Ara-C also called cytosine arabinoside, and melphalan. BCNU is given on the first day, Ara-C and VP-16 on the second, third, fourth and fifth days, and melphalan on the sixth day. The infusion of blood stem cells is given through the catheter the day after the last dose of chemotherapy. This is called Day 0. A week later the subject will receive shots under the skin of Neupogen to help the stem cells grow quickly. Three additional doses of rituximab are given weekly starting 2 weeks later. If the subject recovers and is discharged from the hospital before getting all the doses of rituximab, they can receive the remainder in clinic.

Patients will remain in the hospital for approximately 3-4 weeks, and in the Houston area for about 30 days from the infusion of the donor cells. The patient will have blood, urine, bone marrow, and x-ray examinations performed as necessary to monitor the results of treatment. They will have blood tests daily while hospitalized.

As an outpatient, the patient will be monitored to make sure their immune system (system in the body that helps protect the body and fights bacterial, viral and fungal infections) is recovering, and the patient may require additional infusions of immunoglobulins (infection-fighting blood proteins) until the blood protein levels are safe. The patient will also be taking antibiotic pills for about 6 months to prevent infections. They will have x-rays and other diagnostic tests (PET scans) every 6-12 months during the next 5 years to make sure the tumor stays under control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven, relapsed, or refractory CD20+ lymphoma, or HD.
* At least 2e6 CD34+/kg autologous PBSC stored. If patients are non-mobilizers, then at least 2e8 TNC/kg autologous marrow should be stored.
* Patient is not pregnant.
* Zubrod performance status less than or equal to 2.
* Life expectancy is not severely limited by concomitant illness.
* Left ventricular ejection fraction greater than or equal to 50%.
* No uncontrolled arrhythmias or symptomatic cardiac disease.
* FEV1, FVC and DLCO greater than or equal to 50%.
* No symptomatic pulmonary disease.
* Serum creatinine less than or equal to 1.5 mg/dL.
* Serum bilirubin less than or equal to 2X upper limit of normal, SGPT less than or equal to 3X upper limit of normal.
* No evidence of chronic active hepatitis or cirrhosis.
* No effusion or ascites greater than or equal to 1L prior to drainage.
* HIV negative.
* Patient or guardian able to sign informed consent.
* Patients of any age may be enrolled on this protocol.

Exclusion Criteria:

* Anyone not meeting the above criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-06; Primary Completion 2014-08 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Carrum, MD, Principal Investigator — Associate Professor; Director-Adult Outpatient Clinic
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituxan+BEAM: Autologous Stem Cell Transplant: Ara-C, VP-16, BCNU, Melphalan, Rituxan and Stem Cells BEAM Conditioning.
  Melphalan: Given on Day -1
  Melphalan is administered according to the current SOP.
  Ara-C: 200 mg/m2 IB BID given on Days -5, -4, -3, -2
  VP-16: 200 mg/m2 IV BID given on Days -5, -4, -3, -2
  BCNU: BCNU 300 mg/m2 IV given on Day -6
  Rituxan: 375 mg/m2 IB given on Days -6, +14, +21, +28
  Stem Cells: Stem cells given on Day 0
Period: Overall Study
Arm/Group | Rituxan+BEAM: Autologous Stem Cell Transplant
Started | 75
Completed | 28
Not Completed | 47
Not completed — Additional treatment | 3
Not completed — Progressive disease | 5
Not completed — Relapse | 20
Not completed — Death | 6
Not completed — Lost to Follow-up | 2
Not completed — Ongoing | 11

BASELINE CHARACTERISTICS:
Arm/Group | Rituxan+BEAM: Autologous Stem Cell Transplant
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 53 [14 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 43
Disease at diagnosis [Number; unit: participants]
  Hodgkin's Disease | 25
  Non-Hodgkin's Lymphoma | 50

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Disease-free survival at 12 months post-transplant in patients with Hodgkin's disease or non-Hodgkin's lymphomas
Time Frame: 12 months post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participant
Groups:
- BEAM + R: Autologous Stem Cell Transplant: Ara-C, VP-16, BCNU, Melphalan, Rituxan and Stem Cells BEAM Conditioning.
  Melphalan: Given on Day -1
  Melphalan is administered according to the current SOP.
  Ara-C: 200 mg/m2 IB BID given on Days -5, -4, -3, -2
  VP-16: 200 mg/m2 IV BID given on Days -5, -4, -3, -2
  BCNU: BCNU 300 mg/m2 IV given on Day -6
  Rituxan: 375 mg/m2 IB given on Days -6, +14, +21, +28
  Stem Cells: Stem cells given on Day 0
Arm/Group | BEAM + R: Autologous Stem Cell Transplant
Number analyzed (Participants) | 75
percentage of participant
  All patients | 76 [65 to 84]
  Hodgkin's Disease | 88 [67 to 96]
  Non-Hodgkin's Lymphomas | 70 [55 to 81]

2. Secondary Outcome: Median Days to Neutrophil Engraftment
Description: Neutrophil engraftment was recorded as the first day that absolute neutrophil counts (ANC) exceeds 0.5 X 10^9/L for three consecutive readings.
Time Frame: 30 days post-transplant
Population: All of the participants enrolled in the study engrafted.
Measure: Median (Full Range); unit: days
Arm/Group | BEAM + R: Autologous Stem Cell Transplant
Number analyzed (Participants) | 75
days | 11 [9 to 23]

3. Secondary Outcome: Number of Participants With Overall Best Response Achieved After Transplantation
Description: Response was summarized as complete remission (CR): disappearance of all evidence of disease; partial remission (PR): regression of measurable disease (>=50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses) and no new sites; stable disease (SD): failure to attain CR/PR/PD; relapsed disease or progressive disease (PD): any new lesion or increase by >= 50% of previously involved sites from nadir.
Time Frame: 3 months post-transplant
Population: Analysis comprised of all participants who received standard BEAM chemotherapy and adjuvant rituximab while undergoing autologous blood stem cell transplantation for high-risk lymphoma or Hodgkin's disease.
Measure: Number; unit: participants
Arm/Group | BEAM + R: Autologous Stem Cell Transplant
Number analyzed (Participants) | 75
participants
  Complete Remission (CR) | 63
  Partial Remission (PR) | 8
  Stable Disease (SD) | 0
  Relapsed Disease or Progressive Disease (PD) | 4

ADVERSE EVENTS:
Time Frame: Adverse events related to the study drug, rituximab, are reported during the period of 30 days after transplant.
Description: Only related adverse events were collected for this study.
Groups:
- Rituxan+BEAM: Autologous Stem Cell Transplant: Ara-C, VP-16, BCNU, Melphalan, Rituxan and Stem Cells BEAM Conditioning.
  BEAM Conditioning.
  Melphalan: Given on Day -1
  Melphalan is administered according to the current SOP.
  Ara-C: 200 mg/m2 IB BID given on Days -5, -4, -3, -2
  VP-16: 200 mg/m2 IV BID given on Days -5, -4, -3, -2
  BCNU: BCNU 300 mg/m2 IV given on Day -6
  Rituxan: 375 mg/m2 IB given on Days -6, +14, +21, +28
  Stem Cells: Stem cells given on Day 0
Arm/Group | Rituxan+BEAM: Autologous Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 1/75
Other Adverse Events (participants affected / at risk) | 2/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituxan+BEAM: Autologous Stem Cell Transplant (N=75)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1) — Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituxan+BEAM: Autologous Stem Cell Transplant (N=75)
Cardiovascular/ General - Other (Cardiac disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Pain - Other (General disorders) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes